CLINICAL TRIAL: NCT00710502
Title: Transvaginal Natural Orifice Translumenal and Endoscopic Surgery (NOTES) Cholecystectomy vs. Laparoscopic Cholecystectomy: Phase I/II Clinical Trial
Brief Title: Transvaginal NOTES Cholecystectomy: Phase I/II Mexico Clinical Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidad Juárez del Estado de Durango (Other)
Collaborators: Hospital Universitario La Paz (Other)
Responsible Party: Homero Rivas MD, Hospital de la Paz
Organization: North Texas Veterans Healthcare System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05626
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Cholelithiasis
Keywords: Transvaginal; NOTES; Cholecystectomy; Laparoscopic
MeSH Terms: conditions — Cholelithiasis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Transvaginal NOTES Cholecystectomy (Phase 1)
  Interventions: Procedure: Transvaginal NOTES cholecystectomy
- 2 (Active Comparator): Laparoscopic Cholecystectomy (Phase 2)
  Interventions: Procedure: Laparoscopic cholecystectomy
- 3 (Experimental): Transvaginal NOTES cholecystectomy (Phase 2)
  Interventions: Procedure: Transvaginal NOTES cholecystectomy

INTERVENTIONS:
Procedure: Transvaginal NOTES cholecystectomy — Under general anesthesia, patients will undergo Transvaginal NOTES cholecystectomy
  Other Names: NOTES gallbladder removal; NOTES gallbladder surgery
  Arms: 1; 3
Procedure: Laparoscopic cholecystectomy — Under general anesthesia, patients will undergo standard Laparoscopic cholecystectomy
  Other Names: Small incision gallbladder surgery
  Arms: 2

SUMMARY:
Cholecystectomy is one of the most common general surgery procedures performed in the US today and is among top 10 procedures performed in U.S. hospitals annually, and biliary tract disease has been estimated to cost U.S. healthcare $5 billion/year. Laparoscopic cholecystectomy was introduced in the early 1990s and has become the standard surgical approach for the treatment of gallbladder disease. More than 500,000 cholecystectomy procedures are performed in the US every year. Laparoscopic cholecystectomy is now performed as an outpatient basis and is related to a very low complication rate. Laparoscopic cholecystectomy requires the use of multiple trocar incisions.

Natural Orifice Translumenal Endoscopic Surgery(NOTES) is a new type of surgical procedure currently being studied around the world. The idea of NOTES was developed several years ago in response to the concepts that patients would

1. realize the benefits of less invasive surgery by reducing the recovery time,
2. experience less physical discomfort associated with traditional procedures
3. have virtually no visible scarring following this type of surgery.

All of these advantages have spurred research and investigation forward, encouraging physicians and researchers to develop new equipment and techniques to use during NOTES procedures. Although the Natural Orifice Translumenal Endoscopic Surgery approach may hold tremendous potential, there are many issues that need to be addressed before this technique is introduced into clinical care.

The purpose of this study is to determine the safety, feasibility and short-term clinical outcomes (Phase I trial) of transvaginal NOTES cholecystectomy in female patients with symptomatic cholelithiasis and compare it to Laparoscopic Cholecystectomy (Phase II).

Hypothesis 1: Transvaginal NOTES cholecystectomy is safe and feasible in female patients with symptomatic cholelithiasis.

Hypothesis 2: The short term outcomes of Transvaginal NOTES cholecystectomy are comparable to Laparoscopic Cholecystectomy in female patients with symptomatic cholelithiasis.

Aim 1: Determine the safety of Transvaginal NOTES cholecystectomy. Aim 2: Determine the feasibility of Transvaginal NOTES cholecystectomy. Aim 3: Determine the short-term outcomes of Transvaginal NOTES cholecystectomy. Aim 4: Compare the short-term outcomes of Transvaginal NOTES cholecystectomy to Laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Most recently, surgeons and endoscopists have focused on NOTES cholecystectomy. Access to the abdominal cavity to perform NOTES procedures has been obtained by transgastric, transvaginal, transvesical and transrectal approaches. The first successful NOTES procedure in humans was an appendectomy in India. Transvaginal NOTES cholecystectomy has been successfully performed and reported in a handful of cases in the US, Europe and South America. However, to date, there is lack of clinical trials that demonstrate the safety and feasibility of Transvaginal NOTES cholecystectomy in a larger group of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (> 18 years old) female patients residents of Durango Mexico.
2. Patients who undergo elective surgery.
3. Patients with ultrasound documented symptomatic cholelithiasis, gallbladder polyps of biliary dyskinesia.
4. Patients capable of giving written informed consent for the study.

Exclusion Criteria:

1. Patients who have contraindications prohibiting general anesthesia.
2. Pregnancy.
3. Previous abdominal or gynecological procedures.
4. Uncontrollable medical or psychiatric conditions
5. Elderly > 65 y/o.
6. Body Mass Index > 35 mg/kg2.
7. Complicated or acute cholecystitis.
8. Elevation of liver function tests.
9. Acute abdomen.
10. Intra-abdominal abscess.
11. Coagulopathy.
12. Imperforated hymen.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety and Efficacy of Transvaginal NOTES cholecystectomy when compared to Laparoscopic cholecystectomy | 12 months

SECONDARY OUTCOMES:
Short term outcomes of Transvaginal NOTES cholecystectomy when compared to Laparoscopic Cholecystectomy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Homero Rivas, MD, Principal Investigator — Hospital de la Paz
Locations (1):
- Universidad Juarez del Estado de Durango, Mexico, Durango, Durango, Mexico